CLINICAL TRIAL: NCT05664568
Title: Early Bactericidal Activity of Cephalexin and Amoxicillin-clavulanate for Susceptible Tuberculosis - BLAST 1 Trial
Brief Title: The BLAST- 1 Trial - Cephalexin+Amoxicillin-clavulanate for Tuberculosis
Acronym: BLAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Sydney Local Health District (Other)
Collaborators: Centre Of Research Excellence in Tuberculosis Control (Unknown)
Responsible Party: Principal Investigator, Jan-Willem Alffenaar, Professor, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/PID01942
Record Dates: First submitted 2022-11-02; First posted 2022-12-23 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Randomized controlled trial; Early bactericidal activity; Smear-positive TB; Betalactam antibiotics; Cephalosporin; Time to positivity
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Cephalexin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: Randomized-controlled early bactericidal activity trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care TB (Active Comparator): Standard of care treatment for TB (rifampicin, isoniazid, ethambutol and pyrazinamide according to WHO)
  Interventions: Other: Standard of care treatment of tuberculosis
- Cephalexin + amoxicillin-clavulanate (Experimental): Intervention arm: cephalexin 1g thrice daily + amoxicillin-clavulanate 500/125 mg thrice daily.
  Interventions: Drug: Cephalexin; Drug: Amoxicillin-Clavulanate 500 Mg-125 Mg Oral Tablet

INTERVENTIONS:
Drug: Cephalexin — Participants in intervention group will receive a combination of cephalexin and amoxicillin-clavulanate for the first 2 weeks of TB treatment
  Other Names: Keflex
  Arms: Cephalexin + amoxicillin-clavulanate
Drug: Amoxicillin-Clavulanate 500 Mg-125 Mg Oral Tablet — Participants in the intervention group will receive a combination of cephalexin and amoxicillin-clavulanate for the first 2 weeks of TB treatment
  Other Names: Augmentin
  Arms: Cephalexin + amoxicillin-clavulanate
Other: Standard of care treatment of tuberculosis — The control group will be given standard of care treatment of tuberculosis consisting of rifampicin, isoniazid, pyrazinamide and ethambutol
  Other Names: HREZ
  Arms: Standard of care TB

SUMMARY:
The goal of this randomized controlled trial is to study the early bactericidal activity in adult patients with smear-positive pulmonary tuberculosis.

The main question it aims to answer are if cephalexin, in combination with amoxicillin-clavulanate, is effective in the treatment of tuberculosis.

Participants with smear-positive tuberculosis will be randomized to either of two groups:

Intervention group: cephalexin and amoxicillin-clavulanate. Control group: Standard of care TB treatment. The study period is 2 weeks and participants will be asked to submit multiple sputum samples to measure the bacterial sputum load. They will also submit saliva samples for estimation of drug concentrations in the body.

Researchers will compare the intervention group with the control group to see if the trial drugs result in a reduced bacterial sputum load

Overall aim: To study the early bactericidal activity of cephalexin, in combination with amoxicillin-clavulanate, in comparison to standard treatment in patients with active pulmonary tuberculosis during the first 2 weeks of treatment.

Primary aim:

1. To evaluate the early bactericidal activity (measured as 'time to culture positivity') of cephalexin-clavulanate in comparison, to standard TB treatment (rifampicin, isoniazid, pyrazinamide, and ethambutol).

   Secondary aim:
2. To asses safety and tolerability of cephalexin together with amoxicillin-clavulanate.
3. To determine key pharmacokinetic (PK) parameters of cephalexin, especially half-life and drug exposure (maximal concentration; Cmax and area under the concentration versus time curve, AUC).

DETAILED DESCRIPTION:
Given the need for alternative and well-tolerated tuberculosis (TB) treatment options, there is scope to re-assess the potential value of already approved drugs that are known to be safe, cheap and widely available. Cephalexin, in combination with amoxicillin-clavulanate, have shown high in vitro efficacy against the TB bacteria. Both cephalexin and amoxicillin-clavulanate are Therapeutic Goods Administration (TGA) approved and are widely used in Australia for common infections.

In order to compare the bacterial killing effect of cephalexin, in combination with amoxicillin-clavulanate, with current standard of care TB treatment, we will perform an open-label randomized controlled trial.

Eligible and consenting study participants with bacteriologically confirmed sputum-smear positive pulmonary TB will be randomised to an intervention or control arm in a 1:1 ratio (15 patients in each arm) for the two weeks duration of the trial.

* Intervention arm: cephalexin 1g thrice daily + amoxicillin-clavulanate 500/125 mg thrice daily.
* Control arm: standard of care treatment for TB (rifampicin, isoniazid, ethambutol and pyrazinamide) The primary outcome is the fall in bacterial load measured by 'time to positive culture' using the BACTEC MGIT system with automated detection. Multiple sputum samples (10 in total) will be collected during the first 2 weeks of TB treatment. Six saliva samples will be collected after 4 days of treatment, in order to estimate the drug concentrations of cephalexin in the body (intervention arm only).

For a small subset of patients receiving cephalexin (n=5), a more intensive simultaneous blood and saliva sampling will be done in order to calculate the saliva:plasma ratio, in order to facilitate the estimation of plasma drug concentrations from saliva samples.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults (≥18 years)
* ≥40 kg
* Smear-positive patients with active tuberculosis, confirmed by sputum smear, TB PCR and/or GeneXpert.

Exclusion Criteria:

* On TB treatment for >1 day
* Condition affecting ability of an informed consent (i.e. dementia, delirium etc).
* Pregnancy or breast-feeding
* HIV
* Known allergy or sensitivity to any of the study drugs
* Drug-resistant TB (resistance to rifampicin and/or isoniazid)
* Poor general condition or severe infection such that, in the opinion of the investigator at screening, any delay in initiation of definitive TB treatment cannot be tolerated
* TB with concomitant central nervous system and/or cardiac involvement.
* Any condition as determined by physical examination, medical history, laboratory data, or chest x-ray which, in the opinion of the investigator, would interfere with safety or endpoint assessments in the study.
* Use of metformin, probenecid or allopurinol
* Known previous Clostridium difficile infection due to the risk of colitis. (In case no medical records are available, it should be suspected in elderly patients reporting severe gastrointestinal infections in relation to courses of antibiotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to positivity (TTP) | 2 weeks
  Early bactericidal activity measured as fall in time to positivity (TTP)
  1. The primary outcome is fall in bacterial load in sputum, measured as the rate of change in Time to Sputum Culture Positivity (TTP). TTP is the time to a positive culture when sputum samples are incubated in BACTEC MGIT for automated detection of M. tuberculosis. Measuring the fall in bacterial load is standard choice of outcome for studies evaluating the effect (kill) of drug on TB bacteria.

SECONDARY OUTCOMES:
Adverse events | 2 weeks
  Tolerability - frequency, categorization and grade of adverse events according to CTCAE (Common Terminology Criteria for Adverse Events)
Area under the concentration versus time curve (AUC) of cephalexin | 2 weeks
  Estimation of the pharmacokinetic parameter area under the concentration versus time curve (AUC) of cephalexin in saliva.
Cmax of cephalexin | 2 weeks
  Estimation of the pharmacokinetic parameter maximum concentration (Cmax) of cephalexin saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, Professor, Principal Investigator — WSLHD, Department of Pharmacy, Westmead hospital, NSW, Australia
Locations (3):
- Australia (3):
  - Blacktown Hospital, Sydney
  - Royal Prince Alfred Hospital, Sydney
  - Western Sydney Health District, Sydney